CLINICAL TRIAL: NCT04557501
Title: PSMA PET/CT Guided Intensification of Therapy in Patients at Risk of Advanced Prostate Cancer
Acronym: PATRON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Lantheus Medical Imaging (Industry); British Columbia Cancer Agency (Other); London Health Sciences Centre (Other); Princess Margaret Hospital, Canada (Other); Tom Baker Cancer Centre (Other); McMaster University (Other); Institute of Health Economics, Canada (Other); Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.208
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - SOC Treatment (Active Comparator): Participants to receive surgery or radiotherapy (+/- hormone therapy) as planned per SOC.
  Interventions: Other: Control Arm
- Experimental - PSMAiTx (Experimental): Participants undergo PSMA PET/CT prior to treatment, and treated intensified based on image findings.
  Interventions: Diagnostic Test: PSMA PET/CT guided intensification of therapy

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT guided intensification of therapy — PSMA PET/CT prior to treatment.
  Arms: Experimental - PSMAiTx
Other: Control Arm — Control - Treatment without PSMA PET/CT
  Arms: Control - SOC Treatment

SUMMARY:
Through the conduct of a Phase III randomized controlled trial, investigators plan to: 1) determine if PSMA PET/CT guided intensification of radiotherapy or surgery improves cancer outcomes compared to conventional imaging-guided therapy in patients at risk of advanced disease, 2) evaluate its impact on toxicity and quality of life, and 3) measure the cost-effectiveness of the PSMA PET/CT guided approach.

Participants with high-risk prostate cancer planned for curative-intent standard-of-care radiotherapy or surgery, or with biochemical failure after radical prostatectomy planned for salvage radiotherapy will be enrolled over 3 years (n=776). Those randomized to the investigational arm will have PSMA PET/CT prior to therapy. Based on the imaging results, treating physicians will intensify radiotherapy or surgery unless widely metastatic disease is found, in which case systemic therapy will be intensified.

DETAILED DESCRIPTION:
PSMA PET/CT, particularly with the new generation [18F]DCFPyL radiotracer, has substantially improved our ability to detect sites of prostate cancer compared with conventional imaging alone. When combined with innovative radiotherapeutic and surgical techniques that can now safely target and ablate such disease sites, next generation imaging is now poised to transform the therapeutic paradigm for patients at risk of advanced cancer.

Investigators postulate that intensification of radiotherapy or surgery based on the results of PSMA PET/CT will improve cancer control outcomes in a cost-effective manner, with minimal toxicity, and an overall improvement in quality of life in the longer term.

Investigators expect to show that PSMA PET/CT will have a direct and profound impact on radiotherapy and surgery practice, translating to improved failure-free survival outcomes in patients at risk of advanced prostate cancer. The subset of patients potentially impacted is broad, including patients recurring after prostatectomy and newly presenting patients with high-risk features. Although PSMA PET/CT is increasingly making its way into clinical practice around the world, Canadian provinces will need to make an informed decision of whether to fund this imaging for our patients. The high-level evidence gathered in this trial is desperately needed to assess the impact on patient outcomes and, in doing so, justify broad access and reimbursement for patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of adenocarcinoma of the prostate planned for curative-intent standard-of-care radiotherapy (primary or salvage post prostatectomy) or radical prostatectomy with lymph node dissection.
* Age ≥ 18
* High risk of regional or distant metastases as defined by any of:
* Newly diagnosed and untreated prostate cancer with CAPRA score 6-10, or stage cN1.
* Prior history of radical prostatectomy and biochemical failure (PSA>0.1ng/mL).
* Patients must provide study-specific informed consent prior to study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Active or prior androgen deprivation therapy (except 5-alpha reductase inhibitor) terminated < 12 months prior to enrollment.
* Prior or planned PSMA PET/CT scan outside of this clinical trial.
* Charlson Comorbidity Index > 5 (see Appendix 2).
* Prior curative intent treatment for prostate cancer with local therapy other than surgery (primary radiotherapy or ablative therapies)
* Evidence of extra-pelvic nodal disease (M1a) on conventional imaging (if performed)
* Evidence of metastatic disease (M1b bone, M1c viscera/soft tissue) on conventional imaging (if performed)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To determine if PSMA PET/CT guided intensification of therapy is superior to standard of care (SOC) therapy as measured by improved failure-free survival (FFS). | 5 years

SECONDARY OUTCOMES:
Rates of toxicity (CTCAE) | 5 years
Time to subsequent next-line therapy | 5 years
Quality of Life (EPIC 26) | 5 years
New lesion detection yield (on PSMA PET/CT) | 3 years
Impact of PMSA PET/CT on RT or surgical management (rate of treatment intensification) | 3 years
Cost-effectiveness (EQ5D5L) | 5 years

CONTACTS AND LOCATIONS:
Locations (19):
- Canada (19):
  - BC Cancer Kelowna, Kelowna, British Columbia
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - St-Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital de la Cité de la Santé, Laval, Quebec
  - Charles Lemoyne Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CHU de Québec, Québec, Quebec
  - CHUS, Sherbrooke, Quebec
  - Tom Baker Cancer Center, Calgary
  - Cross Cancer Institute, Edmonton
  - CHUM, Montreal
  - Jewish General Hospital, Montreal
  - Windsor Regional Cancer Centre, Windsor
  - Cancer Care Manitoba, Winnipeg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menard C, Young S, Zukotynski K, Hamilton RJ, Benard F, Yip S, McCabe C, Saad F, Brundage M, Nitulescu R, Bauman G. PSMA PET/CT guided intensification of therapy in patients at risk of advanced prostate cancer (PATRON): a pragmatic phase III randomized controlled trial. BMC Cancer. 2022 Mar 8;22(1):251. doi: 10.1186/s12885-022-09283-z. PMID 35260100